CLINICAL TRIAL: NCT04172103
Title: The Association Between the Duration of Acute Kidney Injury and New-onset Chronic Kidney Disease After Cardiac or Thoracic Aortic Surgery: a Retrospective Observational Cohort Study
Brief Title: The Association Between the Duration of Acute Kidney Injury and New-onset Chronic Kidney Disease After Cardiac or Thoracic Aortic Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1909-115-1066
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease, Stage 3; Chronic Kidney Disease, Stage 5; Cardiac Surgery; Thoracic Aortic Surgery
Keywords: acute kidney injury; chronic kidney disease; cardiac surgery; thoracic aortic surgery
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to evaluate the association between the duration and stage of acute kidney injury (AKI) and the development of chronic kidney disease during postoperative three years in patients undergoing cardiac or thoracic aortic surgery.

DETAILED DESCRIPTION:
Postoperative acute kidney injury (AKI) has been investigated as an important contributor to postoperative morbidity and mortality after cardiovascular surgery. Also, temporary worsening of renal function after aortic surgery is associated with higher long-term mortality. Although the associations between AKI and chronic kidney disease (CKD) in medical or other surgical settings were reported, only a few studies evaluated this relationship in patients undergoing cardiac surgery. More specifically, the association of the severity or duration of AKI with the risk of the development of new-onset CKD after cardiac surgery has not been clearly elucidated.

It would be important to find predictors of the long-term renal function or risk factors for the development of CKD after cardiac surgery because postoperative management of high-risk patients to develop long-term renal dysfunction may prevent further deterioration in renal function and improve patient prognosis.

The investigators aimed to evaluate (1) the long-term renal function after cardiac surgery and (2) the association between the duration and stage of acute kidney injury (AKI) and the development of chronic kidney disease during postoperative three years in patients undergoing cardiac or thoracic aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent cardiac or thoracic aortic surgery under cardiopulmonary bypass at Seoul National University Hospital between 2008 and 2017

Exclusion Criteria:

* Those with off-pump coronary artery bypass
* Missing baseline serum creatinine
* Missing postoperative serum creatinine values of more than three among seven postoperative days
* Preoperative baseline chronic kidney disease with estimated glomerular filtration rate <60 ml/min/1.73m2

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort of the adult patients who underwent cardiac or thoracic aortic surgery under cardiopulmonary bypass at Seoul National University Hospital between 2008 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 2009 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
new-onset chronic kidney disease stage 3 or higher or mortality | during 3 years after surgery
  development of new-onset chronic kidney disease stage 3 or higher or all-cause mortality developed during 3 years after surgery. The new-onset chronic kidney disease was defined by at least two estimated Glomerular Filtration Rate values <60 ml/min/1.73 m2 separated by an interval of at least three months.

SECONDARY OUTCOMES:
new-onset chronic kidney disease stage 3 or higher or mortality | during 1 year after surgery
  development of new-onset chronic kidney disease stage 3 or higher or all-cause mortality developed during 1 year after surgery
new-onset chronic kidney disease stage 3 or higher or mortality | during 2 years after surgery
  development of new-onset chronic kidney disease stage 3 or higher or all-cause mortality developed during 2 years after surgery
Length of postoperative hospital stay | during one month after surgery
  Length of postoperative hospital stay
Length of postoperative intensive care unit stay | during one month after surgery
  Length of postoperative intensive care unit stay
intra-aortic balloon pulsation insertion | during surgery and postoperative one week
  intra-aortic balloon pulsation insertion
Reopen for surgical bleeding | during one month after surgery
  Reopen for surgical bleeding
Respiratory complication | during one month after surgery
  a composite outcome including postoperative atelectasis, pneumonia, pulmonary edema, pleural effusion and pneumothorax
in-hospital mortality | during one month after surgery
  all-cause mortality during hospital stay
Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2 | at three months after surgery
  Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2
Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2 | at one year after surgery
  Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2
Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2 | at two years after surgery
  Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2
Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2 | at three years after surgery
  Incidence of estimated Glomerular Filtration Rate <60 mL/min/1.73m2
Dependence on the regular hemodialysis | at three years after surgery
  Dependence on the regular hemodialysis
estimated Glomerular Filtration Rate | at three months after surgery
  estimated Glomerular Filtration Rate
estimated Glomerular Filtration Rate | at one year after surgery
  estimated Glomerular Filtration Rate
estimated Glomerular Filtration Rate | at two years after surgery
  estimated Glomerular Filtration Rate
estimated Glomerular Filtration Rate | at three years after surgery
  estimated Glomerular Filtration Rate

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Bellomo R. Cardiac surgery-associated acute kidney injury: risk factors, pathophysiology and treatment. Nat Rev Nephrol. 2017 Nov;13(11):697-711. doi: 10.1038/nrneph.2017.119. Epub 2017 Sep 4. PMID 28869251
- [Background] Chawla LS, Eggers PW, Star RA, Kimmel PL. Acute kidney injury and chronic kidney disease as interconnected syndromes. N Engl J Med. 2014 Jul 3;371(1):58-66. doi: 10.1056/NEJMra1214243. No abstract available. PMID 24988558
- See also: Statistical analysis plan — https://doi.org/10.6084/m9.figshare.10326734.v1